CLINICAL TRIAL: NCT05636410
Title: Ultrasound Assessment of the Larynx and Trachea in the Neonatal Period
Status: Completed | Type: Observational
Sponsor: Princess Anna Mazowiecka Hospital, Warsaw, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: LARYNXUS
Record Dates: First submitted 2022-06-13; First posted 2022-12-05 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2023-05

CONDITIONS: Larynx; Trachea
Keywords: larynx; trachea; newborn; ultrasound; anatomy
MeSH Terms: conditions — Laryngeal Diseases; Tracheal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Larynx and trachea ultrasound — After meeting enrolment criteria the larynx and trachea ultrasound will be performed at 32 and 42 weeks of gestation.

SUMMARY:
Diseases of the larynx and trachea are a heterogenous group of disorders. Witch may include congenital anatomical disorders, neoplastic changes, vocal cord paralysis of varied aetiology or narrowing of the larynx associated with long-term intubation. The multitude of disorders of these organs necessitates the continuing search for diagnostic methods which will not only provide answers to clinical questions but will also be safe and with the least level of interference with the wellbeing of the patient, which is of particular importance in the neonate.

In recent decades only a few studies have been reported which described the ultrasound anatomy of the larynx prior to and following intubation or that of the mobility of the vocal cords. To date, no standards have been published concerning the size of the structures of the larynx and trachea or the mobility of the vocal cords on ultrasound examination in the neonate. Additionally, there are no recommendations which include ultrasound examination as a reliable component of the diagnosis of congenital disorders of the larynx or other diseases of this organ.

Ultrasound is a non-invasive, repeatable and safe diagnostic method, which has recently, thanks the development of technology, provided for the very accurate imaging of even small structures, as well as their assessment on dynamic examination. Furthermore, the easy availability of this examination may in the future contribute to the early diagnosis of diseases of the larynx and trachea without the need to prolong neonatal hospitalization or anaesthesia.

In addition, the use of neural networks to analyse the ultrasound images obtained will provide for the development of algorithms which could become an irreplaceable tool, not only in the diagnosis of the disorders described, but also in predicating disorders affecting their further development or functional disorders in infancy.

DETAILED DESCRIPTION:
Diseases of the larynx and trachea are a heterogenous group of disorders. Witch may include congenital anatomical disorders, neoplastic changes, vocal cord paralysis of varied aetiology or narrowing of the larynx associated with long-term intubation. The multitude of disorders of these organs necessitates the continuing search for diagnostic methods which will not only provide answers to clinical questions but will also be safe and with the least level of interference with the wellbeing of the patient, which is of particular importance in the neonate.

Diagnosis of diseases of the larynx and trachea in the neonate and infant is mainly based on endoscopy, magnetic resonance imaging and computer tomography. These investigations are invasive and not infrequently require anaesthetising the patient.

In recent decades only a few studies have been reported which described the ultrasound anatomy of the larynx prior to and following intubation or that of the mobility of the vocal cords. These studies involved small groups of subjects and were performed using lower quality ultrasound devices which did not provide for unequivocal conclusions to be drawn. To date, no standards have been published concerning the size of the structures of the larynx and trachea or the mobility of the vocal cords on ultrasound examination in the neonate. Additionally, there are no recommendations which include ultrasound examination as a reliable component of the diagnosis of congenital disorders of the larynx or other diseases of this organ.

Ultrasound is a non-invasive, repeatable and safe diagnostic method, which has recently, thanks the development of technology, provided for the very accurate imaging of even small structures, as well as their assessment on dynamic examination. Furthermore, the easy availability of this examination may in the future contribute to the early diagnosis of diseases of the larynx and trachea without the need to prolong neonatal hospitalization or anaesthesia.

In addition, the use of neural networks to analyse the ultrasound images obtained will provide for the development of algorithms which could become an irreplaceable tool, not only in the diagnosis of the disorders described, but also in predicating disorders affecting their further development or functional disorders in infancy.

The aim of the study is the accurate description of the ultrasound anatomy of the larynx and trachea and to establish reference ranges for the size of individual structures of the larynx and trachea in the neonatal population.

The study also aims to develop a universal method of ultrasound assessment of the mobility of the vocal cords on dynamic examination and to determine a rule for predicting the expected size of the laryngeal and tracheal structures in relation to anthropometric measurements.

Furthermore, the aim of the study is to promote the use of a non-invasive examination, such as ultrasonography, in the diagnosis of diseases of the larynx and trachea in the youngest patients.

Additionally, the study will be conducted in order to develop artificial intelligence algorithms based on artificial neural networks.

ELIGIBILITY:
Inclusion Criteria:

- gestational age ≥32 weeks

Exclusion Criteria:

* gestational age < 32 weeks,
* presence of significant congenital anomalies,
* intubated neonate,
* unstable neonate.

Ages: 0 Days to 28 Days | Sex: All
Age Groups: Child
Study Population: We plan to recruit all consecutive infants borned at 32 and 42 weeks of gestation.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Larynx and trachea anatomy description. | Through study completion, an average of 2 years
  The aim of the study is the accurate description of the ultrasound anatomy of the larynx and trachea and establishment of reference ranges for the size of individual structures of the larynx and trachea in the neonatal population.
Ultrasound assessment of the mobility of the vocal cords | Through study completion, an average of 2 years
  The study also aims to develop a universal method of ultrasound assessment of the mobility of the vocal cords on dynamic examination and to determine a rule for predicting the expected size of the laryngeal and tracheal structures in relation to anthropometric measurements.
Artificial intelligence algorithms based on artificial neural networks | Through study completion, an average of 2 years
  The study will be conducted in order to develop artificial intelligence algorithms based on artificial neural networks.

CONTACTS AND LOCATIONS:
Overall Officials: Renata Bokiniec, M. D, Study Chair — Dr hab. n. med.
Locations (2):
- Poland (2):
  - Department of Neonatology, Ujastek Medical Center, Krakow, Lesser Poland Voivodeship
  - Department of Neonatology and Neonatal Intensive Care Warsaw Medical University, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be available, after deidentication. The study protocol will also be available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: June 2022 - December 2022
Access Criteria: Documents will be accessible to anyone who provides a methodologically sound proposal immediately following publication with no end date.

REFERENCES:
- [Background] Ongkasuwan J, Ocampo E, Tran B. Laryngeal ultrasound and vocal fold movement in the pediatric cardiovascular intensive care unit. Laryngoscope. 2017 Jan;127(1):167-172. doi: 10.1002/lary.26051. Epub 2016 Apr 23. PMID 27107409
- [Background] Beale T, Twigg VM, Horta M, Morley S. High-Resolution Laryngeal US: Imaging Technique, Normal Anatomy, and Spectrum of Disease. Radiographics. 2020 May-Jun;40(3):775-790. doi: 10.1148/rg.2020190160. PMID 32364882
- [Background] Singh S, Jindal P, Ramakrishnan P, Raghuvanshi S. Prediction of endotracheal tube size in children by predicting subglottic diameter using ultrasonographic measurement versus traditional formulas. Saudi J Anaesth. 2019 Apr-Jun;13(2):93-99. doi: 10.4103/sja.SJA_390_18. PMID 31007653
- [Background] Physical status: the use and interpretation of anthropometry. Report of a WHO Expert Committee. World Health Organ Tech Rep Ser. 1995;854:1-452. PMID 8594834
- [Derived] Paprocki LP, Migda B, Bokiniec R. Ultrasound assessment of larynx and trachea in the neonatal period - analysis of correlations and percentile charts. J Ultrason. 2025 Dec 31;25(103):20250034. doi: 10.15557/jou.2025.0034. eCollection 2025 Oct. PMID 41555932
- [Derived] Paprocki L, Migda B, Bokiniec R. Ultrasound assessment of larynx and trachea in the neonatal period-reference values. Eur Radiol. 2026 Jan;36(1):423-432. doi: 10.1007/s00330-025-11794-9. Epub 2025 Jul 10. PMID 40634702
- [Derived] Paprocki L, Migda B, Bokiniec R. Ultrasound Assessment of Larynx and Trachea in the Neonatal Period, Examination Standard with Predictive Values-Study Protocol. Diagnostics (Basel). 2023 Apr 28;13(9):1578. doi: 10.3390/diagnostics13091578. PMID 37174969